CLINICAL TRIAL: NCT03328689
Title: Community Based Secondary Prevention of Back Pain Flare-ups (Back2LiveWell): a Randomized Controlled Trial
Brief Title: Back2LiveWell: Community Based Prevention of Back Pain Flare-ups
Acronym: Back2LiveWel
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: McMaster University (Other)
Collaborators: Macquarie University, Australia (Other); University of Alberta (Other); Universidade Federal do Ceara (Other)
Responsible Party: Principal Investigator, Luciana Macedo, Assistant Professor, McMaster University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: Back2LiveWell2017
Record Dates: First submitted 2017-10-23; First posted 2017-11-01 (Actual); Last update posted 2020-02-21 (Actual); Status verified 2020-02

CONDITIONS: Low Back Pain, Recurrent; Low Back Pain
Keywords: prevention; exercise; randomized controlled trial; physical activity
MeSH Terms: conditions — Low Back Pain; Motor Activity

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Masking Description: Given that this is an exercise study blinding of participants and those delivering the exercise program will not be possible. Outcome measures will be collected by an investigator not aware of treatment allocation, but most outcome measures will be self-reported and thus, true assessor blinding will no be possible. All statistical analysis will be conducted by a blinded investigator.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Physical activity in the community (Experimental): The physical activity program will include an individualized exercise program delivered in community exercise facility plus education..
  Interventions: Other: Physical activity program
- Control group standard care (Active Comparator): Participants from the control group will receive no additional intervention other than being encouraged to continue with their physiotherapists or chiropractor recommendation which will often include recommendation to keep activity, home exercise programs and advice to engage in physical activity.
  Interventions: Other: Control group standard care

INTERVENTIONS:
Other: Physical activity program — This arm will begin with PT assessment. Following this, participants will meet with a specialist who will design an individualized physical activity program. Classes will include warm up, 40 minutes of individualized exercises and a cool down that will include back pain specific exercises including core strengthening. The first 4 weeks of exercise will include a 30-minute education program. Education comprise information on back pain, efficient use of the back during daily activities, self-management, self-efficacy and pain neurophysiology. Classes will run for a 12-week period. Participants will be encouraged to attend the exercise facility at least 3 times a week. An activity monitor will be provided to all participants. We will use group classes to facilitate the development of social support.
  Arms: Physical activity in the community
Other: Control group standard care — Participants from the control group will receive usual care which will often include recommendation to keep activity, home exercise programs and advice to engage in physical activity.
  Participants in the control group will also receive and activity monitor for collection of physical activity data. This activity monitor may also be used for positive feedback and activity reinforcement
  Arms: Control group standard care

SUMMARY:
The primary objective of this study is to compare the effectiveness and cost-effectiveness of an individualized group based exercise and education program supported in the community to a control group of usual care in preventing back pain flare-ups and to mitigate the negative consequences of subsequent episodes if they occur.

DETAILED DESCRIPTION:
Secondary objectives are to:

• To compare the effectiveness of the two interventions in preventing an activity-limiting LBP flare up at 12 and 24 months.

Secondary objectives are to:

* To compare the effectiveness of the interventions in mitigating the negative consequences of LBP.
* To evaluate the cost-effectiveness of the interventions in preventing activity-limiting LBP flare-up.
* To identify subgroups of individuals that may best respond to each one of the two interventions.

Exploratory objectives include:

* evaluate the fluctuating nature of back pain using a smart phone application to collect pain measures once a week for 1 year (trajectories will also be evaluated to compare between group effects)
* assess adherence to physical activity using activity monitors.
* evaluate the relationship between activity levels and flare-ups as a method for understanding pain triggers and impact of activity pacing.

ELIGIBILITY:
Inclusion criteria:

Participants will be included if they meet the following criteria

* Have been discharged <3 months from physiotherapy, chiropractic or osteopathic care following a course of treatment for LBP (pain in the area between the 12th rib and buttock crease)
* Have non-specific LBP which is pain not attributed to a specific diagnosis such as sciatica, ankylosing spondylitis, vertebral fracture, etc.
* Non-specific LBP sometimes called mechanical LBP accounts for ~85% of LBP diagnosis.
* Between 18 and 80 years of age

Exclusion criteria:

Participants will be excluded if they meet the following criteria:

* Ongoing high pain intensity, defined as pain intensity of 6 or more on a 0-10 point scale. The cut off of 6/10 is used in the literature to dichotomise low/moderate to high pain intensity.
* Co-morbidity preventing participation in physical activity evaluated using the Physical Activity Readiness Questionnaire (PAR-Q) from the American College of Sports Medicine guidelines
* Inadequate English to complete outcome measures
* Currently participating in an exercise program similar to the one we will evaluate.
* History of spine surgery

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 17 (Actual)
Dates: Start 2018-11-25 (Actual); Primary Completion 2019-12-31 (Actual); Study Completion 2019-12-31 (Actual)

PRIMARY OUTCOMES:
Activity limiting flare-up | 12 months
  * flare-up is an increase in pain levels of greater than or equal to 3 on a 0-10 numeric pain scale. The LBP international consensus on minimal important change in pain is 2 on a 0-10 scale and thus a change of 3 is likely be clinically important.15
  * activity-limiting LBP will be measured using an adaptation of the item PI9 of the PROMIS item bank. (How much did LBP interfere with your day to day activities?) A score of 3 or greater (representing somewhat impact) on a 1-5 scale will be considered as activity limitation.
  Participants will fit the criteria for activity-limiting flare-up if pain increases at least 3 points AND pain is identified to be limiting on the PI9 as described above.
  Flare-up will be collected once a week for 1 year

SECONDARY OUTCOMES:
Activity limiting flare-up | 3 and 6 months
  * flare-up is an increase in pain levels of greater than or equal to 3 on a 0-10 numeric pain scale. The LBP international consensus on minimal important change in pain is 2 on a 0-10 scale and thus a change of 3 is likely be clinically important.15
  * activity-limiting LBP will be measured using an adaptation of the item PI9 of the PROMIS item bank. (How much did LBP interfere with your day to day activities?) A score of 3 or greater (representing somewhat impact) on a 1-5 scale will be considered as activity limitation.
  Participants will fit the criteria for activity-limiting flare-up if pain increases at least 3 points AND pain is identified to be limiting on the PI9 as described above.
  Flare-up will be collected once a week for 1 year
Personal Impact of low back pain | 3, 6, 12 months
  the outcome combines 9 items from the Patient Reported Outcome Measurement Information System (PROMIS) short form and covers the domains of pain intensity, pain interference with normal activities and functional status widely recommended in consensus documents on outcome measures for back pain
Pain intensity _NRS pain | 3, 6, 12 months
  Pain intensity over the last week will be measured using a numeric rating scale 0-10 where 0 is not pain and 10 is worse pain
Disability | 3, 6, 12 months
  Roland Morris Disability Questionnaire is a scale from 0-24 assessing pain related disability where 0 is no disability and 24 is significant disability
Function | 3, 6, 12 months
  Patient Specific Functional Scale is a self reported scale assessing function on a scale from 0-10 where 0 is not able to perform the activity and 10 is able without pain
Health related Quality of Life: EQ-5D-5L | 3, 6, 12 months (0-100)
  EQ-5D-5L
Physical activity questionnaire | 3, 6, 12 months
  IPAQ_short form
Physical activity level | 3, 6, 12 months
  Activity level measured using Garmin physical activity monitor

CONTACTS AND LOCATIONS:
Overall Officials: Luciana Macedo, PhD, Principal Investigator — McMaster University
Locations (1):
- YMCA Hamilton, Hamilton, Ontario, Canada

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Macedo LG, Richardson J, Battie MC, Hancock M, Kwan M, Hladysh G, Zhuo L. Back to living well: community-based management of low back pain: a feasibility study. Pilot Feasibility Stud. 2021 Jun 24;7(1):134. doi: 10.1186/s40814-021-00863-7. PMID 34167584